CLINICAL TRIAL: NCT01410890
Title: A Phase 3/4 Prospective Study to Characterize the Pharmacokinetics of Alglucosidase Alfa in Patients With Pompe Disease
Brief Title: Pharmacokinetics of Alglucosidase Alfa in Patients With Pompe Disease
Acronym: PAPAYA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AGLU07710; 2010-022231-11 (EudraCT Number); MSC12790 (Other: Sanofi)
Record Dates: First submitted 2011-08-02; First posted 2011-08-05 (Estimated); Results first posted 2021-06-11 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Pompe Disease; Glycogen Storage Disease Type II (GSD II)
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alglucosidase alfa (Experimental): Participants received intravenous (IV) infusion of Alglucosidase alfa 20 milligrams per kilogram (mg/kg) body weight on Day 1. Infusion was administered at an initial rate of approximately 1 milligram per kilogram per hour (mg/kg/hr) with allowed rate increased of 2 mg/kg/hr every 30 minutes, if there were no signs of infusion-associated reactions (IARs), until a maximum rate of approximately 7 mg/kg/hr was reached.
  Interventions: Biological: alglucosidase alfa

INTERVENTIONS:
Biological: alglucosidase alfa — Intravenous (IV) infusion of 20mg/kg body weight every other week (qow)
  Other Names: Lumizyme

SUMMARY:
* The primary objective of this study was to characterize the pharmacokinetics (PK) of alglucosidase alfa manufactured at the 4000 L scale in participants who had a confirmed diagnosis of Pompe disease.
* A secondary objective of this study was to evaluate and explore the relationship between anti-recombinant human acid alpha-glucosidase antibody titers and the PK of alglucosidase alfa.

DETAILED DESCRIPTION:
The total study duration per participant was 4 to 8 weeks that consisted of a screening period (from 2 days to 4 weeks), treatment visit (1 day), and a follow up call (greater than or equal to 30 days). Two participants enrolled prior to protocol amendment 2 (dated 17 December 2015), which changed the study to single-dose, and were treated for 26 weeks, with a 4-week follow up.

ELIGIBILITY:
Inclusion Criteria:

A participant was to meet all of the following criteria to be eligible for this study:

* The participant and/or the participant's parent/legal guardian was willing and able to provide signed informed consent.
* The participant had a confirmed acid alpha-glucosidase (GAA) enzyme deficiency from skin, blood, or muscle tissue and/or 2 confirmed GAA gene mutations.
* Infant and toddler Pompe disease participants could be included in the study only under condition (minimal body weight) that the trial-related blood loss (including any losses in the maneuver) would not exceed 3 percent (%) of the total blood volume during a period of 4 weeks and would not exceed 1 % at any single time.
* The participant, if female and of childbearing potential, must have had a negative pregnancy test (urine beta-human chorionic gonadotropin) at screening. Note: All female participants of childbearing potential and sexually mature males must have agreed to use a medically accepted method of contraception throughout the study.
* For participants previously treated with alglucosidase alfa the participant had received alglucosidase alfa for at least 6 months.

Exclusion Criteria:

A participant who met any of the following criteria was excluded from this study:

* The participant was participating in another clinical study using an investigational product.
* The participant, in the opinion of the Investigator, was unable to adhere to the requirements of the study.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-11-03 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (12):
- United States (4):
  - Investigational Site Number 840008, Valhalla, New York
  - Investigational Site Number 840007, Cincinnati, Ohio
  - Investigational Site Number 840005, Salt Lake City, Utah
  - Investigational Site Number 840003, Fairfax, Virginia
- Investigational Site Number 1028, Sofia, Bulgaria
- India (2):
  - Investigational Site Number 356001, New Delhi
  - Investigational Site Number 356002, Vellore
- Russia (2):
  - Investigational Site Number 643001, Moscow
  - Investigational Site Number 643002, Moscow
- Investigational Site Number 804001, Kiev, Ukraine
- United Kingdom (2):
  - Investigational Site Number 826003, Birmingham
  - Investigational Site Number 826002, Salford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Nicolas X, Hurbin F, Periquet M, Richards S, Sensinger C, Welch K, An Haack K. Pharmacokinetics of Alglucosidase Alfa Manufactured at the 4000-L Scale in Participants with Pompe Disease: A Phase 3/4 Open-Label Study. Clin Pharmacol Drug Dev. 2023 Dec;12(12):1185-1193. doi: 10.1002/cpdd.1314. Epub 2023 Sep 13. PMID 37705424

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 12 sites in 6 countries. A total of 27 participants were screened between 03-Nov-2014 and 23-Sep-2020, of whom 6 participants were screen failures and 21 participants were enrolled in the study.
Pre-assignment Details: Out of 21 participants, 1 participant signed the informed consent, but due to health status did not continue in the study to the treatment visit.
Groups:
- Alglucosidase Alfa: <18 Years: Participants with less than (<) 18 years of age received intravenous (IV) infusion of Alglucosidase alfa 20 milligram per kilogram (mg/kg) body weight on Day 1. Infusion was administered at an initial rate of approximately 1 milligrams per kilogram per hour (mg/kg/hr) with allowed rate increased of 2 mg/kg/hr every 30 minutes, if there were no signs of infusion-associated reactions (IARs), until a maximum rate of approximately 7 mg/kg/hr was reached.
- Alglucosidase Alfa: >=18 Years: Participants with greater than or equal to (>=) 18 years of age received IV infusion of Alglucosidase alfa 20 mg/kg body weight on Day 1. Infusion was administered at an initial rate of approximately 1 mg/kg/hr with allowed rate increased of 2 mg/kg/hr every 30 minutes, if there were no signs of IARs, until a maximum rate of approximately 7 mg/kg/hr was reached.
Period: Overall Study
Arm/Group | Alglucosidase Alfa: <18 Years | Alglucosidase Alfa: >=18 Years
Started | 10 | 11
Treated | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Full analysis set (FAS) that included all participants who received any amount of alglucosidase alfa.
Groups:
- Alglucosidase Alfa: <18 Years: Participants with <18 years of age received IV infusion of Alglucosidase alfa 20 mg/kg body weight on Day 1. Infusion was administered at an initial rate of approximately 1 mg/kg/hr with allowed rate increased of 2 mg/kg/hr every 30 minutes, if there were no signs of IARs, until a maximum rate of approximately 7 mg/kg/hr was reached.
- Alglucosidase Alfa: >=18 Years: Participants with >=18 years of age received IV infusion of Alglucosidase alfa 20 mg/kg body weight on Day 1. Infusion was administered at an initial rate of approximately 1 mg/kg/hr with allowed rate increased of 2 mg/kg/hr every 30 minutes, if there were no signs of IARs, until a maximum rate of approximately 7 mg/kg/hr was reached.
- Total: Total of all reporting groups
Arm/Group | Alglucosidase Alfa: <18 Years | Alglucosidase Alfa: >=18 Years | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.1 (3.95) | 41.8 (12.44) | 23.4 (20.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 5 | 8 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 6 | 8 | 14
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 9 | 14
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Anti-Recombinant Human Acid Alpha-Glucosidase (rhGAA) Immunoglobulin G (IgG) Antibody Status [Count of Participants; unit: Participants] — Positive antibody status indicated presence of anti-rhGAA IgG antibodies and negative antibody status indicated absence of anti-rhGAA IgG antibodies.
  Participants
    Positive | 3 | 4 | 7
    Negative | 6 | 6 | 12
    Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Plasma Concentration (Cmax) of Alglucosidase Alfa
Description: Cmax was defined as maximum observed plasma concentration.
Time Frame: Pre-dose and at 1, 2, 4, 8, 12, and 24 hours Post-dose on Day 1
Population: Analysis was performed on all participants who received any amount of alglucosidase alfa.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Alglucosidase Alfa: <18 Years | Alglucosidase Alfa: >=18 Years
Number analyzed (Participants) | 10 | 10
nanograms per milliliter (ng/mL) | 204000 (94600) | 307000 (143000)

2. Primary Outcome: Pharmacokinetics: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Alglucosidase Alfa
Description: Tmax was defined as time to reach maximum observed plasma concentration.
Time Frame: Pre-dose and at 1, 2, 4, 8, 12, and 24 hours Post-dose on Day 1
Population: Analysis was performed on all participants who received any amount of alglucosidase alfa.
Measure: Median (Full Range); unit: hours
Arm/Group | Alglucosidase Alfa: <18 Years | Alglucosidase Alfa: >=18 Years
Number analyzed (Participants) | 10 | 10
hours | 4.23 [1.92 to 6.42] | 3.85 [1.42 to 5.33]

3. Primary Outcome: Pharmacokinetics: Area Under the Plasma Concentration-Time Curve (AUC) of Alglucosidase Alfa
Description: AUC was defined as area under the plasma concentration-time curve from time 0 to 24 hours post-dose.
Time Frame: Pre-dose and at 1, 2, 4, 8, 12, and 24 hours Post-dose on Day 1
Population: Analysis was performed on all participants who received any amount of alglucosidase alfa.
Measure: Mean (Standard Deviation); unit: hours per nanograms per milliliter
Arm/Group | Alglucosidase Alfa: <18 Years | Alglucosidase Alfa: >=18 Years
Number analyzed (Participants) | 10 | 10
hours per nanograms per milliliter | 1110000 (753000) | 1890000 (969000)

4. Primary Outcome: Pharmacokinetics: Area Under the Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-last) of Alglucosidase Alfa
Description: AUC0-last was defined as area under the concentration-time curve from time 0 to the time of the last quantifiable concentration.
Time Frame: Pre-dose and at 1, 2, 4, 8, 12, and 24 hours Post-dose on Day 1
Population: Analysis was performed on all participants who received any amount of alglucosidase alfa.
Measure: Mean (Standard Deviation); unit: hours per nanograms per milliliter
Arm/Group | Alglucosidase Alfa: <18 Years | Alglucosidase Alfa: >=18 Years
Number analyzed (Participants) | 10 | 10
hours per nanograms per milliliter | 1040000 (590000) | 1840000 (901000)

5. Primary Outcome: Pharmacokinetics: Terminal Elimination Half-life (T1/2) of Alglucosidase Alfa
Description: T1/2 was defined as the time taken by drug to reduce to half of its initial plasma concentration.
Time Frame: Pre-dose and at 1, 2, 4, 8, 12, and 24 hours Post-dose on Day 1
Population: Analysis was performed on all participants who received any amount of alglucosidase alfa.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Alglucosidase Alfa: <18 Years | Alglucosidase Alfa: >=18 Years
Number analyzed (Participants) | 10 | 10
hours | 5.43 (3.82) | 3.84 (0.801)

6. Primary Outcome: Pharmacokinetics: Total Systemic Clearance (CL) of Alglucosidase Alfa
Description: CL of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: Pre-dose and at 1, 2, 4, 8, 12, and 24 hours Post-dose on Day 1
Population: Analysis was performed on all participants who received any amount of alglucosidase alfa.
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Alglucosidase Alfa: <18 Years | Alglucosidase Alfa: >=18 Years
Number analyzed (Participants) | 10 | 10
Liters per hour | 0.529 (0.613) | 1.26 (1.24)

7. Primary Outcome: Pharmacokinetics: Volume of Distribution at Steady State (Vss) of Alglucosidase Alfa
Description: Volume of distribution (Vd) is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vss is the apparent volume of distribution at steady-state.
Time Frame: Pre-dose and at 1, 2, 4, 8, 12, and 24 hours Post-dose on Day 1
Population: Analysis was performed on all participants who received any amount of alglucosidase alfa.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Alglucosidase Alfa: <18 Years | Alglucosidase Alfa: >=18 Years
Number analyzed (Participants) | 10 | 10
Liters | 2.35 (2.02) | 5.59 (3.72)

8. Secondary Outcome: Pharmacokinetics: Maximum Observed Plasma Concentration of Alglucosidase Alfa in Anti-Recombinant Human Acid Alpha-Glucosidase Antibody Positive and Negative Participants
Description: Cmax was defined as maximum observed plasma concentration.
Time Frame: Pre-dose and at 1, 2, 4, 8, 12, and 24 hours Post-dose on Day 1
Population: Analysis was performed on FAS that included all participants who received any amount of alglucosidase alfa. Here, overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Anti-rhGAA Antibody Negative Participants: Participants with negative anti-rhGAA IgG antibody status at Baseline received IV infusion of Alglucosidase alfa 20 mg/kg body weight on Day 1. Infusion was administered at an initial rate of approximately 1 mg/kg/hr with allowed rate increased of 2 mg/kg/hr every 30 minutes, if there were no signs of IARs, until a maximum rate of approximately 7 mg/kg/hr was reached.
- Anti-rhGAA Antibody Positive Participants: Participants with positive anti-rhGAA IgG antibody status at Baseline received IV infusion of Alglucosidase alfa 20 mg/kg body weight on Day 1. Infusion was administered at an initial rate of approximately 1 mg/kg/hr with allowed rate increased of 2 mg/kg/hr every 30 minutes, if there were no signs of IARs, until a maximum rate of approximately 7 mg/kg/hr was reached.
Arm/Group | Anti-rhGAA Antibody Negative Participants | Anti-rhGAA Antibody Positive Participants
Number analyzed (Participants) | 12 | 7
ng/mL | 256000 (121000) | 262000 (160000)

9. Secondary Outcome: Pharmacokinetics: Time to Reach Maximum Observed Plasma Concentration in Anti-rhGAA Antibody Positive and Negative Participants
Description: Tmax was defined as time to reach maximum observed plasma concentration.
Time Frame: Pre-dose and at 1, 2, 4, 8, 12, and 24 hours Post-dose on Day 1
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | Anti-rhGAA Antibody Negative Participants | Anti-rhGAA Antibody Positive Participants
Number analyzed (Participants) | 12 | 7
hours | 3.94 [1.92 to 5.27] | 4.33 [1.42 to 6.42]

10. Secondary Outcome: Pharmacokinetics: Terminal Elimination Half-life of Alglucosidase Alfa in Anti-rhGAA Antibody Positive and Negative Participants
Description: T1/2 was defined as the time taken by drug to reduce to half of its initial plasma concentration.
Time Frame: Pre-dose and at 1, 2, 4, 8, 12, and 24 hours Post-dose on Day 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Anti-rhGAA Antibody Negative Participants | Anti-rhGAA Antibody Positive Participants
Number analyzed (Participants) | 12 | 7
hours | 4.68 (2.95) | 4.79 (2.93)

11. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration of Alglucosidase Alfa in Anti-rhGAA Antibody Positive and Negative Participants
Description: AUC0-last was defined as area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration.
Time Frame: Pre-dose and at 1, 2, 4, 8, 12, and 24 hours Post-dose on Day 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours per nanograms per milliliter
Arm/Group | Anti-rhGAA Antibody Negative Participants | Anti-rhGAA Antibody Positive Participants
Number analyzed (Participants) | 12 | 7
hours per nanograms per milliliter | 1410000 (865000) | 1610000 (86800)

12. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-time Curve From Time 0 and Extrapolated to Infinite Time (AUC0-inf) in Anti-rhGAA Antibody Positive and Negative Participants
Description: AUC0-inf was defined as area under the concentration-time curve from time 0 extrapolated to infinite time.
Time Frame: Pre-dose and at 1, 2, 4, 8, 12, and 24 hours Post-dose on Day 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours per nanograms per milliliter
Arm/Group | Anti-rhGAA Antibody Negative Participants | Anti-rhGAA Antibody Positive Participants
Number analyzed (Participants) | 12 | 7
hours per nanograms per milliliter | 1450000 (941000) | 1700000 (985000)

13. Secondary Outcome: Pharmacokinetics: Total Systemic Clearance in Anti-rhGAA Antibody Positive and Negative Participants
Description: CL of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: Pre-dose and at 1, 2, 4, 8, 12, and 24 hours Post-dose on Day 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Anti-rhGAA Antibody Negative Participants | Anti-rhGAA Antibody Positive Participants
Number analyzed (Participants) | 12 | 7
Liters per hour | 0.765 (0.518) | 1.21 (1.60)

14. Secondary Outcome: Pharmacokinetics: Volume of Distribution in Anti-rhGAA Antibody Positive and Negative Participants
Description: Vd is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vss is the apparent volume of distribution at steady-state.
Time Frame: Pre-dose and at 1, 2, 4, 8, 12, and 24 hours Post-dose on Day 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Anti-rhGAA Antibody Negative Participants | Anti-rhGAA Antibody Positive Participants
Number analyzed (Participants) | 12 | 7
Liters | 5.82 (6.49) | 7.26 (9.16)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to Week 4.
Description: Reported AEs and deaths were treatment-emergent (TEAEs) that developed/worsened in grade/became serious during 'TEAE period' (i.e., from signature of the informed consent form up to Week 4. Analysis was performed on FAS that included all participants who received any amount of alglucosidase alfa.
Arm/Group | Alglucosidase Alfa: <18 Years | Alglucosidase Alfa: >=18 Years
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alglucosidase Alfa: <18 Years (N=10) | Alglucosidase Alfa: >=18 Years (N=10)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alglucosidase Alfa: <18 Years (N=10) | Alglucosidase Alfa: >=18 Years (N=10)
Fungal Skin Infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Blood Pressure Increased (Investigations) | 1 (1) | 0 (0)
Body Temperature Increased (Investigations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2016-07-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT01410890/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-23): https://cdn.clinicaltrials.gov/large-docs/90/NCT01410890/SAP_001.pdf